CLINICAL TRIAL: NCT07091708
Title: EFFECT OF ELECTROACUPUNCTURE ON COMPLEX REGIONAL PAIN SYNDROME IN PATIENTS WITH STROKE: A RANDOMIZED CONTROLLED TRIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eyad Mohamed Fathy, Demonstator, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1534998
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Other)
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture

SUMMARY:
Complex regional pain syndrome (CRPS) is a condition marked by pain that may occur spontaneously or in response to stimuli, often disproportionate to the initial injury.(Chae, 2010). In post-stroke complex regional pain syndrome, patients often have simultaneous shoulder and wrist pain. Symptoms may include edema, increased warmth in the hand, and limited in upper extremity joints. (Yu, 2009).The significance of post-stroke complex regional pain syndrome (CRPS) lies not only in its profound impact on pain perception but also in its broader effects on patients' quality of life.(de mos et al.,2007) Managing complex regional pain syndrome involves a multidisciplinary approach with key physical therapy elements like elevation, massage, range of motion exercises, strengthening, and sensory re-education.(Sethy et al., 2017). Electrotherapy modalities include transcutaneous electrical nerve stimulation. (Palmer, 2015). This includes heat treatments like ultrasound, hot and cold packs, and fluidotherapy

DETAILED DESCRIPTION:
In this sense,acupuncture, presents a viable alternative to opioid analgesics for pain relief, offering effective treatment without the risk of dependency. one specific technique, electroacupuncture (ea), enhances traditional acupuncture by applying a small electric current between pairs of needles. research indicates that ea may alleviate pain by activating various bioactive chemicals, engaging multiple mechanisms at the peripheral, spinal, and supraspinal levels. this makes electroacupuncture a promising option for individuals seeking non-addictive pain management solutions.( zhang r, et al 2014).

ELIGIBILITY:
Inclusion Criteria:

* 1. The study involved forty patients male and female aged between 45 and 65 years. 2. A confirmed diagnosis of complex regional pain syndrome through clinical assessment by neurologist using The Budapest criteria for diagnosis of CRPS (Choi et al ., 2013

Exclusion Criteria:

* 1. Pre-existing history of hand problems and shoulder dysfunction prior to experiencing a stroke . 2. Those with an overactive sympathetic system from alternative causes eg.congestive heart failure,chronic kidney disease(Reynolds & Minic, 2023) 8 3. individuals with significant musculoskeletal disorders such as rheumatoid arthritis or metabolic disorders including diabetes 4. Pregnancy

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 5 min
  Visual analogue scale (VAS) is valuable tool for assessing the intensity and frequency of symptoms, particularly pain.